CLINICAL TRIAL: NCT06218446
Title: Transgender Caregivers' and Patients' Representations of Parenthood as Part of a Fertility Preservation Pathway
Acronym: TransFert
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230413; 2023-A00509-36 (Other: IDRCB ANSM)
Record Dates: First submitted 2023-12-19; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Transgenderism; Fertility Issues
Keywords: Transidentity; Preservation of fertility; Parenthood; Representations; Reproductive health
MeSH Terms: conditions — Transsexualism; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
- Care team

SUMMARY:
This research aims to understand the impact of fertility preservation consultation on transgender patients' projection and how the possibility of preserving gametes influences transgender people's transition paths, parenthood projects and health and health of transgender people through qualitative interviews.

This research will also study the representations of members of medical and reproductive biology teams the possible use of stored gametes, and how these representations influence their clinical practice.

clinical practice. To answer the research question, we plan to include 30 patients who have consulted for fertility preservation at the at the CECOS of the Tenon hospital, located in the 20th arrondissement of Paris, and 20 members of the center's healthcare team.

care team.

DETAILED DESCRIPTION:
Since the 2016 law, transgender people no longer need to provide "irreversible and medical proof of a physical transformation" in order to carry out a sex change at the Civil Registry, which puts an end to systematic sterilization and opens up the possibility of a hormonal-only transition. Yet hormonal treatments can have an impact on the fertility of transgender people, compromising a subsequent project for parenthood.

The Reproductive Biology department at Tenon, where the research will take place, now offers self-conservation of female and male gametes before hormone replacement treatments are introduced, or during a therapeutic window. Fertility preservation in transgender women relies primarily on sperm self-preservation. For transgender men, fertility preservation relies on cryopreservation of mature oocytes after ovarian stimulation.

In addition to assessing the psychic impact of care in order to prevent potential deleterious effects, psycho-sexological consultation offers an opportunity to express the desire for a child, a desire often inhibited for a long time, as well as information on the possibilities of reuse.

When it comes to research around the issue of fertility preservation for transgender people, there is often talk of problems concerning access to this care: the discriminatory practices of certain centers that refuse transgender people, the lack of training in transidentity issues for care teams, etc. The coercive weight of the law seems to be enough to evade the issue by moving it into the realm of legislation. And yet, in our clinical experience, the question of gamete reuse is a subject that merits research to determine the obstacles and levers for both caregivers and patients.

ELIGIBILITY:
Inclusion Criteria:

* Any transgender person undergoing fertility preservation in the department
* Any member of the reproductive biology and medicine services team
* Aged 18 and over, with or without children
* Informed and having signed consent to participate in the research project

Exclusion Criteria:

* No social security
* Persons under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For patient : transgender patients consulting as part of a fertility preservation course For care teams : care teams from the biology and reproductive medicine department
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients surveyed who developed or modified a gamete-use project following the fertility preservation consultation. | Up to 2 months
  To understand the impact of the fertility preservation consultation on transgender patients' projection in terms of parenthood.

SECONDARY OUTCOMES:
number of caregivers who raise the issue of gamete reuse during their consultations. | Up to 2 months
  To study the way in which caregivers perceive the possible use of preserved gametes, and how these perceptions influence their clinical practice.
number of members of the healthcare team who have changed their practice since the service began accepting transgender patients | Up to 2 months
  To study the way in which caregivers perceive the possible use of preserved gametes, and how these perceptions influence their clinical practice.
  criteria:
Number of patients who have developed a parental project following consultation with the psychologist. | Up to 2 months
Number of patients who are aware of the law and their rights in terms of gamete preservation and use | Up to 2 months
Number of patients who have modified the temporality of their transition (medical and/or administrative) because of their preservation path and/or their desire for parenthood. | Up to 2 months
Number of patients for whom the intention to preserve their gametes is experienced as improving their transition path. | Up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Emilie MOREAU, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CECOS / service de Biologie de la Reproduction Hôpital Tenon, Paris, France

IPD SHARING:
Plan to Share IPD: No